CLINICAL TRIAL: NCT02892955
Title: Multi-Center Study of MagLev Technology in Patients Undergoing MCS Therapy With HeartMate 3™ Continued Access Protocol: Post-Approval Continued Follow-up
Brief Title: MOMENTUM 3 Continued Access Protocol
Acronym: MOMENTUM 3 CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOMENTUM 3 CAP
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Results first posted 2022-03-03 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Advanced Refractory Left Ventricular Heart Failure
Keywords: Heart Failure; LVAS; Ventricular Dysfunction; Cardiomyopathy; Heart Disease; Cardiovascular Disease; Heart-assist devices; Thoratec Corporation
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HeartMate 3 LVAS (HM3 LVAS) (Experimental): The study was a single-arm, prospective, multi-center, study for continued evaluation of safety and clinical performance of the HM3 LVAS.
  Interventions: Device: HeartMate 3 LVAS

INTERVENTIONS:
Device: HeartMate 3 LVAS — Implantation of HeartMate 3 LVAD to evaluate safety and clinical performance of the HM3 LVAS for the treatment of advanced, refractory, left ventricular heart failure following completion of enrollment in the MOMENTUM 3 IDE Study.

SUMMARY:
The objective of the study is to continue to evaluate safety and clinical performance of the HM3 LVAS for the treatment of advanced, refractory, left ventricular heart failure following completion of enrollment in the the MOMENTUM 3 IDE Study.

DETAILED DESCRIPTION:
Enrollment in the CAP cohort ended shortly after approval for the long-term indication was received from the FDA in October 2018. As a condition of approval, all patients enrolled in the CAP cohort were to complete the 2-year follow-up to fulfil a post-approval study requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal representative has signed Informed Consent Form (ICF)
2. Age ≥ 18 years
3. BSA ≥ 1.2 m2
4. NYHA Class III with dyspnea upon mild physical activity or NYHA Class IV
5. LVEF ≤ 25%
6. a) Inotrope dependent OR b) CI < 2.2 L/min/m2, while not on inotropes and subjects must also meet one of the following:

   * On optimal medical management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and are failing to respond
   * Advanced heart failure for at least 14 days AND dependent on intra-aortic balloon pump (IABP) for at least 7 days,
7. Females of child bearing age must agree to use adequate contraception

Exclusion Criteria:

1. Etiology of HF due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, or restrictive cardiomyopathy
2. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator
3. Existence of ongoing mechanical circulatory support (MCS) other than IABP
4. Positive pregnancy test if of childbearing potential
5. Presence of mechanical aortic cardiac valve that will not be either converted to a bioprosthesis or oversewn at the time of LVAD implant
6. History of any organ transplant
7. Platelet count < 100,000 x 103/L (< 100,000/ml)
8. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management
9. History of confirmed, untreated Abdominal Aortic Aneurysm (AAA) > 5 cm in diameter within 6 months of enrollment
10. Presence of an active, uncontrolled infection
11. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy that the investigator will require based upon the patients' health status
12. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:

    * An INR ≥ 2.0 not due to anticoagulation therapy
    * Total bilirubin > 43 umol/L (2.5 mg/dl), shock liver, or biopsy proven liver cirrhosis
    * History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, and FEV1 <50% predicted
    * Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention
    * History of stroke within 90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 80%) uncorrected carotid artery stenosis
    * Serum Creatinine ≥ 221 umol/L (2.5 mg/dl) or the need for chronic renal replacement therapy
    * Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration
13. Patient has moderate to severe aortic insufficiency without plans for correction during pump implant
14. Pre albumin < 150 mg/L (15mg/dL) or Albumin < 30g/L (3 g/dL) (if only one available); pre albumin < 150 mg/L (15mg/dL) and Albumin < 30g/L (3 g/dL) (if both available)
15. Planned Bi-VAD support prior to enrollment
16. Patient has known hypo or hyper coagulable states such as disseminated intravascular coagulation and heparin induced thrombocytopenia
17. Participation in any other clinical investigation that is likely to confound study results or affect the study
18. Any condition other than HF that could limit survival to less than 24 months
19. Patients actively listed for heart transplant (this exclusion applies only after commercial approval of the HM3 for short-term use)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1685 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elena Brett, Study Director — Abbott Medical Devices
Locations (69):
- United States (69):
  - Baptist Health Medical Center - Little Rock, Little Rock, Arkansas
  - Cedars Sinai Medical Center, Beverly Hills, California
  - University of California, San Diego, La Jolla, California
  - Sutter Memorial Hospital, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Hospital @ University of Florida, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health/Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky - Saha Cardiovascular Research Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins Unversity Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Hershey, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas West Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Memorial Hermann Health Systems, Houston, Texas
  - Methodist Houston, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Netuka I, Sood P, Pya Y, Zimpfer D, Krabatsch T, Garbade J, Rao V, Morshuis M, Marasco S, Beyersdorf F, Damme L, Schmitto JD. Fully Magnetically Levitated Left Ventricular Assist System for Treating Advanced HF: A Multicenter Study. J Am Coll Cardiol. 2015 Dec 15;66(23):2579-2589. doi: 10.1016/j.jacc.2015.09.083. PMID 26670056
- [Background] Uriel N, Adatya S, Mehra MR. Evolution in Mechanical Circulatory Support: Are We at the Precipice of a Disruptive Innovation? J Am Coll Cardiol. 2015 Dec 15;66(23):2590-2593. doi: 10.1016/j.jacc.2015.10.028. No abstract available. PMID 26670057
- [Background] Schmitto JD, Hanke JS, Rojas SV, Avsar M, Haverich A. First implantation in man of a new magnetically levitated left ventricular assist device (HeartMate III). J Heart Lung Transplant. 2015 Jun;34(6):858-60. doi: 10.1016/j.healun.2015.03.001. Epub 2015 Mar 7. No abstract available. PMID 25920932
- [Background] Netuka I, Kvasnicka T, Kvasnicka J, Hrachovinova I, Ivak P, Marecek F, Bilkova J, Malikova I, Jancova M, Maly J, Sood P, Sundareswaran KS, Connors JM, Mehra MR. Evaluation of von Willebrand factor with a fully magnetically levitated centrifugal continuous-flow left ventricular assist device in advanced heart failure. J Heart Lung Transplant. 2016 Jul;35(7):860-7. doi: 10.1016/j.healun.2016.05.019. Epub 2016 May 31. PMID 27435529
- [Background] Bourque K, Cotter C, Dague C, Harjes D, Dur O, Duhamel J, Spink K, Walsh K, Burke E. Design Rationale and Preclinical Evaluation of the HeartMate 3 Left Ventricular Assist System for Hemocompatibility. ASAIO J. 2016 Jul-Aug;62(4):375-83. doi: 10.1097/MAT.0000000000000388. PMID 27195742
- [Background] Hanke JS, Haverich A, Schmitto JD. Exchange of a HeartMate II left ventricular assist device with a HeartMate 3 pump. J Heart Lung Transplant. 2016 Jul;35(7):944-6. doi: 10.1016/j.healun.2016.03.013. Epub 2016 Mar 30. No abstract available. PMID 27160494
- [Background] Heatley G, Sood P, Goldstein D, Uriel N, Cleveland J, Middlebrook D, Mehra MR; MOMENTUM 3 Investigators. Clinical trial design and rationale of the Multicenter Study of MagLev Technology in Patients Undergoing Mechanical Circulatory Support Therapy With HeartMate 3 (MOMENTUM 3) investigational device exemption clinical study protocol. J Heart Lung Transplant. 2016 Apr;35(4):528-36. doi: 10.1016/j.healun.2016.01.021. Epub 2016 Jan 30. PMID 27044532
- [Background] Schulz A, Stepanenko A, Krabatsch T. HeartMate 3 implantation via left lateral thoracotomy with outflow graft anastomosis to the descending aorta. J Heart Lung Transplant. 2016 May;35(5):690-2. doi: 10.1016/j.healun.2016.01.004. Epub 2016 Jan 15. No abstract available. PMID 26944673
- [Background] Stansfield WE, Rao V. HeartMate 3: Facing the challenge of past success. J Thorac Cardiovasc Surg. 2016 Sep;152(3):683-5. doi: 10.1016/j.jtcvs.2016.04.048. Epub 2016 Apr 22. No abstract available. PMID 27210469
- [Background] Takayama H. Did you like Terminator 3 better than Terminator 2? "Rise of machines" with HeartMate 3? J Thorac Cardiovasc Surg. 2016 Sep;152(3):686-7. doi: 10.1016/j.jtcvs.2016.05.044. Epub 2016 Jun 2. No abstract available. PMID 27349284
- [Result] Mehra MR, Cleveland JC Jr, Uriel N, Cowger JA, Hall S, Horstmanshof D, Naka Y, Salerno CT, Chuang J, Williams C, Goldstein DJ; MOMENTUM 3 Investigators. Primary results of long-term outcomes in the MOMENTUM 3 pivotal trial and continued access protocol study phase: a study of 2200 HeartMate 3 left ventricular assist device implants. Eur J Heart Fail. 2021 Aug;23(8):1392-1400. doi: 10.1002/ejhf.2211. Epub 2021 May 18. PMID 33932272
- [Derived] Uriel N, Sayer GT, Elad B, Fried JA, Raikhelkar JK, Lotan D, Goldstein DJ, Jorde UP, Cleveland JC Jr, Mehra MR, Drakos SG, Wood KL, Henderson JD, San Lee F, Kanwar MK, Clerkin KJ. Heart Replacement Therapy in Young Patients: A Comparative Analysis of HeartMate 3 LVAD and Heart Transplant Using MOMENTUM 3 and UNOS Registry. JACC Heart Fail. 2026 Feb 6:102948. doi: 10.1016/j.jchf.2026.102948. Online ahead of print. PMID 41653179
- [Derived] Sayer G, Ahmed MM, Mehra MR, Gosev I, Vidula H, Devore AD, Horstmanshof DA, Cleveland JC Jr, Stewart GC, Slaughter MS, Mudy K, Wang A, Uriel N. Implantable Cardioverter-Defibrillators and Cardiovascular Resynchronization Therapy with Left Ventricular Assist DevicesA MOMENTUM 3 Trial Analysis. J Card Fail. 2025 Oct;31(10):1548-1557. doi: 10.1016/j.cardfail.2024.12.011. Epub 2025 Jan 22. PMID 39855458
- [Derived] Molina EJ, Ahmed MM, Sheikh FH, Cleveland JC Jr, Goldstein DJ, Uriel NY, Wang A, Revis JJ, Mehra MR. Left Ventricular Dimensions and Clinical Outcomes With a Fully Magnetically Levitated Left Ventricular Assist Device. JACC Heart Fail. 2025 May;13(5):798-811. doi: 10.1016/j.jchf.2024.09.019. Epub 2024 Dec 18. PMID 39708027
- [Derived] Ramu B, Cogswell R, Ravichandran AK, Cleveland J Jr, Mehra MR, Goldstein D, Uriel N, Dirckx N, Ahmed S, Yuzefpolskaya M. Clinical Outcomes With a Fully Magnetically Levitated Left Ventricular Assist Device Among Women and Men. JACC Heart Fail. 2023 Dec;11(12):1692-1704. doi: 10.1016/j.jchf.2023.08.020. Epub 2023 Oct 11. PMID 37831046
- [Derived] Mehra MR, Nayak A, Morris AA, Lanfear DE, Nemeh H, Desai S, Bansal A, Guerrero-Miranda C, Hall S, Cleveland JC Jr, Goldstein DJ, Uriel N, Chen L, Bailey S, Anyanwu A, Heatley G, Chuang J, Estep JD. Prediction of Survival After Implantation of a Fully Magnetically Levitated Left Ventricular Assist Device. JACC Heart Fail. 2022 Dec;10(12):948-959. doi: 10.1016/j.jchf.2022.08.002. Epub 2022 Oct 12. PMID 36456068
- [Derived] Uriel N, Milano C, Agarwal R, Lee S, Cleveland J, Goldstein D, Wang A, Crandall D, Mehra MR. Incidence and clinical correlates of de-novo aortic regurgitation with a fully magnetically levitated left ventricular assist device: a MOMENTUM 3 trial portfolio analysis. Eur J Heart Fail. 2023 Feb;25(2):286-294. doi: 10.1002/ejhf.2746. Epub 2022 Nov 29. PMID 36404406
- [Derived] Vidula H, Takeda K, Estep JD, Silvestry SC, Milano C, Cleveland JC Jr, Goldstein DJ, Uriel N, Kormos RL, Dirckx N, Mehra MR. Hospitalization Patterns and Impact of a Magnetically-Levitated Left Ventricular Assist Device in the MOMENTUM 3 Trial. JACC Heart Fail. 2022 Jul;10(7):470-481. doi: 10.1016/j.jchf.2022.03.007. Epub 2022 Jun 8. PMID 35772857
- [Derived] Sheikh FH, Ravichandran AK, Goldstein DJ, Agarwal R, Ransom J, Bansal A, Kim G, Cleveland JC, Uriel N, Sheridan BC, Chomsky D, Patel SR, Dirckx N, Franke A, Mehra MR. Impact of Race on Clinical Outcomes After Implantation With a Fully Magnetically Levitated Left Ventricular Assist Device: An Analysis From the MOMENTUM 3 Trial. Circ Heart Fail. 2021 Oct;14(10):e008360. doi: 10.1161/CIRCHEARTFAILURE.120.008360. Epub 2021 Sep 16. PMID 34525837

RESULTS

PARTICIPANT FLOW:
Groups:
- HeartMate 3 LVAS (HM3 LVAS): The study will be a single-arm, prospective, multi-center, study for continued evaluation of safety and clinical performance of the HM3 LVAS.
  HeartMate 3 LVAS: Implantation of HeartMate 3 LVAD to evaluate safety and clinical performance of the HM3 LVAS for the treatment of advanced, refractory, left ventricular heart failure following completion of enrollment in the the MOMENTUM 3 IDE Study.
Period: Overall Study
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Started | 1685
Completed | 1685
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343
  Male | 1342
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants in the "more than one race" category include those who also specified a race other than Asian, Native Hawaiian or Other Pacific Islander, Black or African American, or White race.
  Participants
    American Indian or Alaska Native | 0
    Asian | 19
    Native Hawaiian or Other Pacific Islander | 10
    Black or African American | 466
    White | 1135
    More than one race | 53
    Unknown or Not Reported | 2
INTERMACS Profile [Count of Participants; unit: Participants] — Lower profiles are considered worse. Profile 1 describes patients in critical cardiogenic shock. Profile 2 describes patients with inotrope dependence who show signs of continuing deterioration. Profile 3 describes stable, inotrope dependent patients. Profile 4 describes patients at home on oral therapy with symptoms of congestion at rest. Profile 5 describes exertion intolerant patients who are comfortable at rest. Profile 6 describes exertion limited patients who are comfortable at rest. Profile 7 describes clinically stable patients with reasonable levels of comfortable activity.
  Participants
    1 | 69
    2 | 517
    3 | 843
    4 | 216
    5 | 24
    6 or 7 | 1
    Not provided | 15
Intended Goal of Support [Count of Participants; unit: Participants] — Bridge to recovery: Use of a durable device to allow recovery from chronic cardiac failure. Rescue therapy: Use of a durable device to support resolution from an acute event without major previous cardiac dysfunction. Bridge to transplant: Patient listed for transplant or listed within 24 hours before device implantation. Bridge to candidacy: Patient may be eligible for transplant. Destination therapy: patient definitely not eligible for transplant.
  Participants
    Bridge to Transplant | 173
    Bridge to Candidacy | 233
    Destination Therapy | 1274
    Bridge to Recovery | 4
    Rescue Therapy | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival
Description: Survival at 24 months free of disabling stroke (Modified Rankin Score > 3) or reoperation to replace or remove a malfunctioning device
Time Frame: Subjects will be followed for 24 months or to outcome (transplant, explant, or death), whichever occurs first.
Measure: Count of Participants; unit: Participants
Groups:
- HeartMate 3 LVAS (HM3 LVAS): Patients implanted with HeartMate 3 LVAS and enrolled in the MOMENTUM 3 CAP cohort.
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
Participants | 1320

2. Secondary Outcome: Pump Replacement
Description: Frequency of HeartMate 3 pump replacement at 24 months.
Time Frame: As they occur up to 24 months or to outcome, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
Participants | 20

3. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: Functional status as measured by the Six Minute Walk Test. The Six Minute Walk Test measures the distance a patient is able to walk during 6 minutes without running or jogging.
Time Frame: Baseline, 6 months and 24 months
Population: Analysis population only includes patients still ongoing on LVAD support at the specified time periods who completed the assessment. Patients unable to walk due to heart failure symptoms were assigned a distance of zero.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
meters
  Baseline: number analyzed (Participants) | 1487
  Baseline | 101.3 (160.7)
  6 months: number analyzed (Participants) | 1140
  6 months | 317.2 (163.3)
  24 months: number analyzed (Participants) | 664
  24 months | 305.1 (172.5)

4. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: Functional status as measured by NYHA classification. NYHA class categorizes patients by the severity of their heart failure symptoms. As the class increases, the degree of symptoms is more severe indicating worse functional status. Class I indicates no limitation of physical activity. Class II indicates slight limitation of physical activity. Class IIIA indicates marked limitation of physical activity where less than ordinary physical activity causes fatigue, palpitation, dyspnea, or angina pain. Class IIIB indicates marked limitation of physical activity where mild physical activity causes fatigue, palpitation, dyspnea, or angina pain. Class IV indicates inability to carry on any physical activity without discomfort.
Time Frame: Baseline, 6 months and 24 months
Population: Analysis population only includes patients still ongoing on LVAD support at the specified time periods who completed the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
Participants
  NYHA Class I or II at Baseline: number analyzed (Participants) | 1673
  NYHA Class I or II at Baseline | 0
  Class I or II at 6 Months: number analyzed (Participants) | 1344
  Class I or II at 6 Months | 1046
  Class I or II at 24 Months: number analyzed (Participants) | 949
  Class I or II at 24 Months | 686

5. Secondary Outcome: EuroQol-5D-5L Visual Analogue Scale
Description: Quality of life as measured by the visual analogue scale from the EuroQol-5D-5L questionnaire. The patient rates their current state of health with the visual analogue scale. The scale ranges from 0 to 100. Higher scores indicate a better quality of life.
Time Frame: Baseline, 6 months and 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
score on a scale
  Baseline: number analyzed (Participants) | 1602
  Baseline | 48.3 (25.1)
  6 months: number analyzed (Participants) | 1326
  6 months | 73.9 (18.2)
  24 months: number analyzed (Participants) | 922
  24 months | 72.4 (20.1)

6. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). Scores range from 0 to 100. Higher scores indicate better quality of life and fewer heart failure symptoms.
Time Frame: Baseline, 6 months and 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
Score on a scale
  Baseline: number analyzed (Participants) | 1610
  Baseline | 40.0 (21.6)
  6 months: number analyzed (Participants) | 1325
  6 months | 69.5 (20.0)
  24 months: number analyzed (Participants) | 923
  24 months | 67.3 (21.8)

7. Secondary Outcome: Rehospitalizations
Description: Rate of all cause rehospitalization
Time Frame: From initial discharge to 2 years post-implant
Population: Subjects who were discharged on LVAD support from the implant hospitalization
Measure: Number; unit: events per patient year
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1571
events per patient year | 2.03

8. Secondary Outcome: Adverse Event Rates
Description: Events-per-patient-year (EPPY) for anticipated adverse events as defined in the study protocol
Time Frame: 2 years post-implant
Measure: Number; unit: events per patient year
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
Number analyzed (Participants) | 1685
events per patient year
  Arterial Non-CNS Thromboembolism | 0.01
  Bleeding | 0.71
  Cardiac Arrhythmia | 0.30
  Hepatic Dysfunction | 0.04
  Hypertension | 0.04
  Major Infection | 0.73
  Myocardial Infarction | 0.01
  Stroke | 0.07
  Other Neurological Event | 0.09
  Pericardial Fluid Collection | 0.04
  Psychiatric Episode | 0.07
  Renal Dysfunction | 0.11
  Respiratory Failure | 0.16
  Right Heart Failure | 0.27
  Venous Thromboembolism | 0.03
  Wound Dehiscence | 0.00
  Suspected Device Thrombosis | 0.01
  Hemolysis | 0.00

ADVERSE EVENTS:
Time Frame: 2 years post-implant
Description: Serious adverse events are defined as those adverse events causing death, or congenital abnormality or birth defect, or a life-threatening illness or injury that results in permanent disability, requires hospitalization, or prolongs a hospitalization, and/or requires intervention to prevent permanent injury or damage.
Arm/Group | HeartMate 3 LVAS (HM3 LVAS)
All-Cause Mortality (participants affected / at risk) | 293/1685
Serious Adverse Events (participants affected / at risk) | 1536/1685
Other Adverse Events (participants affected / at risk) | 1050/1685
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HeartMate 3 LVAS (HM3 LVAS) (N=1685)
Protocol defined bleeding (Blood and lymphatic system disorders) | 802 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined hemolysis (Blood and lymphatic system disorders) | 6 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined cardiac arrhythmia (Cardiac disorders) | 473 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined myocardial infarction (Cardiac disorders) | 15 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined pericardial fluid collection (Cardiac disorders) | 96 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined right heart failure (Cardiac disorders) | 541 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined other adverse event (General disorders) | 1084 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined hepatic dysfunction (Hepatobiliary disorders) | 58 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined major infection (Infections and infestations) | 862 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined stroke (Nervous system disorders) | 153 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined other neurological event (Nervous system disorders) | 202 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined suspected device thrombosis (Product Issues) | 18 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined psychiatric episode (Psychiatric disorders) | 73 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined renal dysfunction (Renal and urinary disorders) | 231 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined respiratory failure (Respiratory, thoracic and mediastinal disorders) | 325 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined wound dehiscence (Skin and subcutaneous tissue disorders) | 10 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined arterial non-CNS thromboembolism (Vascular disorders) | 21 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined hypertension (Vascular disorders) | 45 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined venous thromboembolism (Vascular disorders) | 30 — Events categorized based on detailed definition specified in the study protocol.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HeartMate 3 LVAS (HM3 LVAS) (N=1685)
Protocol defined bleeding (Blood and lymphatic system disorders) | 107 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined cardiac arrhythmia (Cardiac disorders) | 135 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined major infection (Infections and infestations) | 267 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined psychiatric episode (Psychiatric disorders) | 94 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined right heart failure (Cardiac disorders) | 107 — Events categorized based on detailed definition specified in the study protocol.
Protocol defined other adverse event (General disorders) | 617 — Events categorized based on detailed definition specified in the study protocol.

LIMITATIONS AND CAVEATS:
This is a single arm study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MOMENTUM 3 studies have a study specific charter that governs the overall publication and presentation policy for all abstracts and manuscripts related to MOMENTUM 3 clinical data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT02892955/Prot_SAP_000.pdf